CLINICAL TRIAL: NCT06165328
Title: The Comparison of Diagnostic Yield Between Routine Computed Tomography and Colonoscope in Detecting Colorectal Tumors in Patients Who at Risk of Colorectal Cancer
Brief Title: The Comparison Between Computed Tomography and Colonoscope in Detecting Colorectal Tumors in Patients With FIT+
Acronym: CTOCOCREC
Status: Recruiting | Type: Observational
Sponsor: Hat Yai Medical Education Center (Other)
Collaborators: HatYai Hospital (Other)
Responsible Party: Principal Investigator, Arunchai Chang, Head of Division of Gastroenterology, Department of Internal Medicine, Hatyai Hospital, Hat Yai Medical Education Center
Other Study IDs: HYH EC 093-66-01
Record Dates: First submitted 2023-12-02; First posted 2023-12-11 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Patients at Risk of Colorectal Cancer
Keywords: colorectal tumor; colorectal cancer; CT scan; colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood for CBC, Coagulogram, BUN, Creatinine, Electrolyte, Iron study, CEA Stool for FIT test pathologic obtained (in case with polyp or malignancy)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort1: Patients with aged more than 50 years and had FIT test +
  Interventions: Diagnostic Test: CT and colonoscopy

INTERVENTIONS:
Diagnostic Test: CT and colonoscopy — All patients were admitted and worked up as inpatient cases. A blood test was obtained and a CT whole abdomen was performed for all patients in the evening. On the next day, all patients were prescribed for bowel preparation in the morning, then subsequently underwent colonoscopy in the afternoon.

SUMMARY:
Colonoscopy is the mainstay modality of choice in colorectal cancer screening worldwide. However, the rate of colonoscopy for colorectal cancer screening is very low (approximately 5-10%) because of the limited local medical resources (such as endoscopists and regional endoscope). This observational diagnostic test study aims to compare the diagnostic yield of routine computed tomography and colonoscopy in detecting colorectal tumors in patients at risk of colorectal cancer (aged more than 50 years and FIT+). The main question[s] it aims to answer are:

1. To compare the diagnostic yield between the routine computed tomography and colonoscopy.
2. To compare the procedure-related adverse events between the routine computed tomography and colonoscopy.

DETAILED DESCRIPTION:
All enrolled patients underwent routine CT scans of whole abdomen, then subsequently under went a colonoscopy on the next day

ELIGIBILITY:
Inclusion Criteria:

1. Fit test +
2. Normal platelet count and normal result of PT, PTT

Exclusion Criteria:

1. pregnancy or lactation
2. uncontrolled Diabetes Mellitus, hypertension, asthma, congestive heart failure
3. recent coronary artery disease within 3 months
4. eGFR lesser than 30 mL/min/1.73m2
5. hemophilia or uncontrolled or uncorrected coagulopathy

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients aged 50-70 years old who underwent FIT test for an indication of colorectal cancer screening as National program of Thailand.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield in diagnosis colorectal tumor | 2 weeks
  Sensitivity, specitivity, accuracy

SECONDARY OUTCOMES:
Procedure-related adverse events | 2 weeks
  Procedure-related adverse events such as, contrast induced nephropathy, contrast allergy, colonoscope-related perforation, post polypectomy bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Arunchai Chang, MD, Principal Investigator — Division of Gastroenetrology, Department of Internal Medicine, Hatyai Hospital
Locations (1):
- Hatyai Hospital, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shaukat A, Levin TR. Current and future colorectal cancer screening strategies. Nat Rev Gastroenterol Hepatol. 2022 Aug;19(8):521-531. doi: 10.1038/s41575-022-00612-y. Epub 2022 May 3. PMID 35505243
- [Result] Wong MCS, Chan FKL. Colorectal cancer screening in middle eastern countries: Current status and future strategies to enhance screening. Saudi J Gastroenterol. 2019 Jan-Feb;25(1):1-2. doi: 10.4103/sjg.SJG_611_18. No abstract available. PMID 30665995
- [Result] Tanaka H, Oka S, Shiotani A, Sugimoto M, Suzuki H, Naito Y, Handa O, Hisamatsu T, Fukudo S, Fujishiro M, Motoya S, Yahagi N, Yamaguchi S, Chan FKL, Lee SY, Li B, Ang TL, Abdullah M, Tablante MC, Prachayakul V, Tanaka S; International Gastrointestinal Consensus Symposium Study Group. Current Status of Diagnosis and Treatment of Colorectal Cancer in Asian Countries: A Questionnaire Survey. Digestion. 2024;105(1):62-68. doi: 10.1159/000531706. Epub 2023 Jul 27. PMID 37497916
- [Result] Ganeshan A, Upponi S, Uberoi R, D'Costa H, Picking C, Bungay H. Minimal-preparation CT colon in detection of colonic cancer, the Oxford experience. Age Ageing. 2007 Jan;36(1):48-52. doi: 10.1093/ageing/afl116. Epub 2006 Nov 17. PMID 17114203
- [Result] Pilleul F, Bansac-Lamblin A, Monneuse O, Dumortier J, Milot L, Valette PJ. Water enema computed tomography: diagnostic tool in suspicion of colorectal tumor. Gastroenterol Clin Biol. 2006 Feb;30(2):231-4. doi: 10.1016/s0399-8320(06)73158-x. PMID 16565655
- [Result] Miller J, Maeda Y, Au S, Gunn F, Porteous L, Pattenden R, MacLean P, Noble CL, Glancy S, Dunlop MG, Din FVN. Short-term outcomes of a COVID-adapted triage pathway for colorectal cancer detection. Colorectal Dis. 2021 Jul;23(7):1639-1648. doi: 10.1111/codi.15618. Epub 2021 Mar 29. PMID 33682302